CLINICAL TRIAL: NCT03942341
Title: The Impact of Alzheimer's Disease on Sleep in Adults With Down Syndrome
Brief Title: Sleep in Adults With Down Syndrome and Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ASD-2019-15
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer's Disease; Obstructive Sleep Apnea; Sleep Disturbances
Keywords: Down syndrome; Alzheimer's disease; obstructive sleep apnea; Polysomnography
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea, Obstructive; Parasomnias; Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult subjects with Down syndrome and Alzheimer Disease: Patients will be included from the 6 centers of the Horizon 21 european consortium. Horizon 21 consortium consists of DS cohorts from Spain (the Down Alzheimer Barcelona Neuroimaging Initiative -DABNI). France (the TriAl 21 at Jérôme Lejeune Institute in Paris), the UK (The LonDowns consortium and Dementia in Down's Syndrome (DiDS) in Cambridge), the Netherlands (the Rotterdam DS cohort) and Germany (AD21 in Munich), with a combined total of more than 1,000 older participants with DS to pool data and bioresources to address current gaps in knowledge about AD in DS.
  All participants will be included after obtaining a written informed consent approved by the ethics committee. A total of 90 DS subjects with AD dementia of both sexes and good general condition will be included. The presence of a family member will be required as well as a sufficient visual and hearing acuity.

SUMMARY:
RATIONALE of the project. Adults with Down syndrome (DS) present severe sleep disorders that are under recognized by caregivers. Aging in DS population increases the prevalence of both Obstructive Sleep Apnea (OSA) and Alzheimer´s disease (AD) dementia at much higher rates than in the general population. AD increases the risk of sleep disturbances and OSA, which in turn worsen cognitive performance and behavioral function.

Our hypothesis is that adults with DS and AD dementia will present a higher prevalence of sleep disorders (sleep disruption, sleep circadian disorders and OSA) than in DS without dementia.

There are no data evaluating nocturnal sleep in adults with DS with AD dementia.

The main objective is to evaluate the prevalence of sleep disturbances in adult subjects with DS and AD dementia, by means of subjective and objectives sleep measures.

DETAILED DESCRIPTION:
Aims To characterize and determine the prevalence of sleep disorders and sleep wake pattern in a large community-based sample of adult subjects with DS and AD dementia and to correlate the results with clinical, cognitive and behavioral features.

OBJECTIVES:

The general objective is to evaluate the impact of AD dementia on sleep in adults with DS.

1. By evaluating the frequency of sleep problems in demented adults with DS through:

   1. Nocturnal sleep by polysomnography (PSG)
   2. Subjective sleep quality (Pittsburg) and daytime Somnolence (Epworth)
   3. Sleep-wake pattern by actimetry
2. By analyzing the association between sleep problems and both age and body mass index (BMI)
3. By analyzing the impact of sleep problems on:

   1. Daytime Somnolence (Epworth, actigraphy)
   2. Diurnal Behavioural disturbances
   3. Neurophysiological performance

   The secondary objective is to compare the sleep data of the DS patients with AD dementia with our sleep data of DS patients without dementia.

   The project is the continuation of our sleep research work in adults with DS. We have performed a community-based cross-sectional study in 54 adults with DS by means of objective and subjective measures, and we found a high prevalence of sleep disorders (Giménez, 2018). In this study, 6 DS patients had AD dementia. Although the sample was very small, our results show that the symptomatic AD-DS group presented a higher apnea hypopnea index (AHI), higher oxygen desaturations (ODI-3%), and higher respiratory arousal index compared to the non demented DS group. The DS group with dementia had also worse sleep efficiency and higher sleep fragmentation.

   METHODS:

   Muliticenter sleep study. Cross-sectional analytical study. The study duration is 24 months. Participants: 90 subjects with DS and AD. Only subjects with mild and moderate mental retardation will be included.

   Variables and method of collection:
   1. Neurological evaluation: Standard visit in which medical and neurological past medical history will be reviewed to apply the inclusion and exclusion criteria.
   2. Neuropsychological evaluation: The neuropsychological battery will be administered by neuropsychologists with experience in the evaluation of DS subjects. The study includes neuropsychological tests that have proven to be sensitive to detect cognitive impairment and is based, in part, from the recommendations of the "Working Group for the Establishment of Criteria for the Diagnosis of Dementia in Individuals with Intellectual Disability." The complete battery has an approximate length of 90 min and consists in:

      - Functional, daily living activities and neuropsychiatric scales.

      - Estimated Intelligence Quotient (IQ): Kaufman Brief Intelligence Test (K-BIT).

      - Global cognition battery adapted to Intellectual Disabilities: CAMDEX-DS, including the structured interview CAMDEX-DS and the cognitive battery CAMCOG-DS.

      - Memory: The Cued Recall Test (CRT) adapted version (Deveny, 2002).
      * Executive function: Cats and dogs test (adaptation of Day-Night Stroop), to measure inhibition capacity and backward digits.
      * Attention: cancellation test.
      * Language: semantic fluency test (animals), 30 items from the Boston Naming Test (BNT).
   3. Sleep evaluation:

   All participants will undergo a full sleep evaluation. This includes a sleep interview with a sleep specialist, and a subjective and objective evaluation of nocturnal sleep and the circadian sleep-wake pattern. Nocturnal sleep will be objectively studied by full video PSG and Sleep/wake pattern will be collected via sleep diaries and actigraphy.

   c.1. Objective sleep measures: Polysomnography (PSG). Sleep recordings will be performed in individual, sound-attenuated, temperature-regulated rooms in sleep units in all groups. Participants will be continuously supervised by qualified technical staff and recorded on video/audio with the use of an infrared camera. PSGs will start at their median bedtime as defined by the prospective diary collection, with a recording time of 8 hours. The morning after the PSG nights, all subjects will complete a subjective questionnaire about their sleep quality in the laboratory. We will compare this questionnaire with their usual reported sleep quality at home.

   All-night video PSG-recordings include: 1) 19 EEG- channels referenced to averaged mastoid electrodes (A1-A2) according to the international 10-20 system; 2) 2 electroculographic channels; and 3) 4 surface electromyographic channels: 2 from the mentalis, one from the right anterior tibialis and one from the left anterior tibialis in lower limbs; and 4) 6 channels to monitor respiratory function: one for oximetry, 2 for oro-nasal airflow using a thermistor and nasal-cannula, 2 to record thoraco-abdominal movements by inductance plethysmography, and a microphone at the suprasternal notch to detect snoring.

   Sleep stages will be visually scored for 30-s epochs according to the guidelines of the American Academy of Sleep Medicine (AASM). Scoring will be performed by an experienced sleep technologist and later reviewed by an accredited sleep specialist.

   Arousals will be defined using AASM criteria. Respiratory variables will include the apnea/hypopnea index (AHI), defined as the sum of all apneas (> 90% reduction in airflow for >10 seconds) and all hypopneas (airflow reduction greater than 30% for at 11 least 10 seconds with an oxygen saturation decrease of approximately 3% or a cortical awakening) per hour of sleep, and mean oxygen saturation during the night (Sp02). Periodic leg movements and abnormal REM sleep behavior disorder will be defined according to the International Criteria of Sleep Disorders.

   c.2. Actigraphy:

   During the week before the PSG, participants will wear an actigraph in the non-dominant arm, a method of monitoring human rest/activity cycles. Variables obtained by actimetry will be analysed in two groups:

   - Activity analysis: variables describing level of activity and light during 24 hours and during all period. Includes average of daily activity during all period, maximum activity times and variance.

   - Sleep analysis: to asses sleep variables derived from actigraphy, bedtime and awake time would be need to know from each subject. These information will be collected through event marker system of the actimeter and from sleep diaries recording.

   c.3. Subjective Sleep Measures (assessed by caregiver): All participants will have a notebook that includes subjective sleep questionnaires and sleep diaries to be completed by the caregivers.

   Sleep questionnaires will include the following scales: the Pittsburgh Sleep Quality Index (PSQI) to assess patients' self-reports of sleep quality; the Epworth Sleepiness Scale (ESS) to evaluate somnolence (with a modification of the last question about the DS person as a passenger in a car while stopped for a few minutes in traffic); and the Berlin Questionnaire (BQ) to identify subjects at risk for the sleep apnea syndrome

   Sleep diary is a daily report of sleep and waking activities over 24-hour periods. The sleep diary reports: bedtime, wake time, how much time taken to fall asleep, how much time spent awake after sleep onset.

   STATISTICAL ANALYSIS:

   Statistical analyses will be performed using SPSS v23 software. Demographics and sleep scores will be compared between groups by means of t tests.

   The statistical threshold is set at 0.05. To assess the differences between the various sleep techniques performed in DS participants, general lineal models (GLM) with one within-subject factor (techniques, 3 levels) will be applied separately to each sleep variable.

   For all variables, results will be pair-compared by means of the t-test. Greenhouse-Geisser correction will be used. The Pearson correlation will be applied to evaluate the relationship between sleep variables.

   STUDY LIMITATIONS The main foreseen limitation for this study it the heterogeneity of the DS population. To try to overcome this difficulty and to facilitate the feasibility of the study, only subjects with mild or mild-moderate mental retardation will be selected.

   ETHICAL ISSUES The study will be carried out in strict accordance with international ethical guidelines for medical research in humans. Researchers are responsible for ensuring that the study is conducted in accordance with standards contained in the Declaration of Helsinki and local regulation. All participants will be included after obtaining a written informed consent (the family member's consent will also be obtained). Before including any subject in the study, the investigator will inform the participant of the objectives, methods and potential risks of the study or any inconvenience this may cause. The studies that will be performed in this project are not part of the routine evaluation of subjects with DS and they have an interest only from a research point of view. To preserve the confidentiality of information, data pertaining to this study will not be included in the conventional medical history, but in a separate file in a protected location.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes with ages over 18 years old with DS.
* Subjects will have to be able to understand and accept the study procedures and sign an informed consent (patient and or guardian).
* Only subjects with mild and moderate mental retardation according to ICD-10criteria (IQ scores> 34).
* Subjects with dementia: subjects with acquired cognitive impairment (assessed by longitudinal neuropsychological tests and/or anamnesis to the family). Absence of comorbid psychiatric disorders (major depressive disorder, bipolar disorder, schizophrenia, autism or behavioral disorders).

Exclusion Criteria:

* Don't meet Inclusion Criteria
* Severe mental retardation
* History of conditions that could affect brain structure or function, such as stroke or traumatic brain injury
* Patients in treatment with CPAP
* New psychoactive drugs in the last three months preceding the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be included after obtaining a written informed consent approved by the ethics committee. A total of 90 DS subjects with AD dementia of both sexes and good general condition will be included. The presence of a family member will be required as well as a sufficient visual and hearing acuity.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | 4 weeks
  The ratio of total sleep time (TST) to time in bed (TIB)

SECONDARY OUTCOMES:
The apnea/hypopnea index (AHI) | 4 weeks
  the sum of all apneas (> 90% reduction in airflow for >10 seconds) and all hypopneas (airflow reduction greater than 30% for at 11 least 10 seconds with an oxygen saturation decrease of approximately 3% or a cortical awakening) per hour of sleep, and mean oxygen saturation during the night (Sp02)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain